CLINICAL TRIAL: NCT01436903
Title: Chances for Success of CavatermTM Surgery as a Function of Uterus Probe Length, a Questionnaire Investigation on 290 Patients
Brief Title: Chances for Success of CavatermTM Surgery as a Function of Uterus Probe Length
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Beda Hartmann, Univ.-Doz. Dr. Mag., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 743/2010
Record Dates: First submitted 2011-08-12; First posted 2011-09-20 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Menorrhagia
Keywords: menorrhagia; dysfunctional uterine bleeding; endometrial ablation; cavatermTM; probe
MeSH Terms: conditions — Menorrhagia; Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thermal Balloon Endometrial Ablation — Thermal Balloon Endometrial Ablation for 10 minutes after curettage
  Other Names: CavatermTM

SUMMARY:
CavatermTM is a second-generation thermal balloon ablation device in the management of menorrhagia. The purpose of this study is to investigate the success (questionnaire) of CavatermTM dependent on uterus probe length, especially corpus probe length, which is measured during surgery.

ELIGIBILITY:
Inclusion Criteria:

* CavatermTM operation because of menorrhagia
* timeframe: January 2006 till August 2009
* older than 29 years and younger than 56 years

Exclusion Criteria:

* pregnancy
* fragmentary filled questionnaire
* more than 1 CavatermTM operation

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Postsurgical change in bleeding patterns dependent on cavum probe length. | Corpus probe length will be measured during surgery, a questionnaire will be sent in September 2010, at least after one postsurgical year.
  Success is defined as a-, hypo- or eumenorrhoea, regular cycle, reduction of dysmenorrhoea.
Postsurgical change in patient satisfaction dependent on cavum probe length. | Corpus probe length will be measured during surgery, a questionnaire will be sent in September 2010, at least after one postsurgical year.
  The questionnaire will ask for satisfaction and recommendation to the best friend.

SECONDARY OUTCOMES:
Postsurgical change in dyspareunia | A questionnaire will be sent in September 2010, at least after one postsurgical year.
  The questionnaire will ask for pre- and postsurgical dyspareunia.
Postsurgical change in Premenstrual Syndrome | A questionnaire will be sent in September 2010, at least after one postsurgical year.
  The questionnaire will ask for pre- and postsurgical Premestrual Syndrome.
Prevention of further gynaecological therapies | A questionnaire will be sent in September 2010, at least after one postsurgical year.
  The questionnaire will ask for postsurgical hysterectomy and further medications.
Improvement of quality of life | A questionnaire will be sent in September 2010, at least after one postsurgical year.
  The questionnaire will ask for postsurgical quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Beda W. Hartmann, Univ.-Doz., Principal Investigator — Medical University of Vienna
Locations (1):
- Landesklinikum Thermenregion Neunkirchen, Neunkirchen, Lower Austria, Austria